CLINICAL TRIAL: NCT03926611
Title: A Multicenter, Randomized, Double-blind, Placebo- Controlled Phase 2b Dose-finding Study to Investigate the Efficacy, Safety and Tolerability of LOU064 in Adult Chronic Spontaneous Urticaria (CSU) Patients Inadequately Controlled by H1-antihistamines
Brief Title: This Was a Dose-finding Study to Evaluate Efficacy and Safety of LOU064 in Patients With CSU Inadequately Controlled by H1-antihistamines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLOU064A2201; 2018-000993-31 (EudraCT Number)
Record Dates: First submitted 2019-04-12; First posted 2019-04-24 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: BTK inhibitor; Urticaria Activity Score; Angioedema Activity Score; CSU
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Intervention Model Description: This was a global Phase 2b multicenter, randomized, double-blind, parallel-group, placebocontrolled study investigating the efficacy, safety and tolerability of 6 dosing groups of oral LOU064 in subjects with inadequately controlled CSU despite treatment with (second generation) H1-antihistamine. Study duration was 18 weeks (2 weeks of screening period; 12 weeks of treatment period and a 4 weeks follow-up period).
  Study had 7 arms: 10 mg LOU064 q.d.; 35 mg LOU064 q.d.; 100 mg LOU064 q.d.; 10 mg LOU064 b.i.d.; 25 mg LOU064 b.i.d.; 100 mg LOU064 b.i.d.; and Placebo
  Throughout study, subjects were treated with a 2nd generation H1-antihistamine at a locally approved licensed posology ("background medication"). Subjects could take an additional second generation H1-antihistamine that was eliminated primarily via renal excretion (e.g. cetirizine, levocetirizine or bilastine) as rescue medication. Eligible subjects could roll over to extension at Wk 12 or Wk 16
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- LOU064 Arm 1 (Experimental): 10 mg LOU064 qd capsule once daily
  Interventions: Drug: LOU064 Arm 1
- LOU064 Arm 2 (Experimental): 35 mg capsule qd LOU064 once daily
  Interventions: Drug: LOU064 Arm 2
- LOU064 Arm 3 (Experimental): 100 mg capsule qd LOU064 once daily
  Interventions: Drug: LOU064 Arm 3
- LOU064 Arm 4 (Experimental): 10 mg capsule LOU064 bid
  Interventions: Drug: LOU064 Arm 4
- LOU064 Arm 5 (Experimental): 25 mg capsule LOU064 bid
  Interventions: Drug: LOU064 Arm 5
- LOU064 Arm 6 (Experimental): 100 mg capsule LOU064 bid
  Interventions: Drug: LOU064 Arm 6
- Placebo Arm (Placebo Comparator): Participants took matching placebo twice daily
  Interventions: Drug: Placebo arm

INTERVENTIONS:
Drug: LOU064 Arm 1 — 10 mg LOU064 orally in the morning (once daily) and matching placebo in the evening from Day 1 to 85
  Arms: LOU064 Arm 1
Drug: LOU064 Arm 2 — 35 mg of LOU064 orally in the morning (once daily) and matching placebo in the evening from Day 1 to 85
  Arms: LOU064 Arm 2
Drug: LOU064 Arm 3 — 100 mg of LOU064 orally in the morning (once daily) and matching placebo in the evening from Day 1 to 85
  Arms: LOU064 Arm 3
Drug: LOU064 Arm 4 — 10mg bid of LOU064 orally, twice daily from Day 1 to 85
  Arms: LOU064 Arm 4
Drug: LOU064 Arm 5 — 25 mg bid of LOU064 orally, twice daily from Day 1 to 85
  Arms: LOU064 Arm 5
Drug: LOU064 Arm 6 — 100 mg bid of LOU064 orally, twice daily from Day 1 to 85
  Arms: LOU064 Arm 6
Drug: Placebo arm — Matching placebo, orally, twice daily from Day 1 to 85
  Arms: Placebo Arm

SUMMARY:
This was a multicenter, randomized, double-blind and placebo-controlled phase 2b dose-finding study to assess the efficacy and safety of LOU064 in adults chronic spontaneous urticaria (CSU) patients inadequately controlled by H1-antihistamines

DETAILED DESCRIPTION:
This was a global Phase 2b multicenter, randomized, double-blind, parallel-group, placebo-controlled study investigating the efficacy, safety and tolerability of six dosing groups of oral LOU064 in subjects with inadequately controlled CSU despite treatment with (second generation) H1-antihistamine. The study comprised of the 7 treatment arms: LOU064 10 mg q.d., LOU064 35 mg q.d., LOU064 100 mg q.d., LOU064 10 mg b.i.d, LOU064 25 mg b.i.d., LOU064 100 mg b.i.d. and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥18 years of age
* CSU diagnosis for ≥ 6 months prior to screening
* Presence of itch and hives for ≥6 consecutive weeks prior to screening in spite of use of non-sedating H1-antihistamines according to local Treatment guidelines during this time period
* UAS7 score (range 0-42) ≥16 and HSS7 score (range 0-21) ≥ 8 during 7 days prior to randomization (Day 1)
* Willing and able to complete an Urticaria Participant Daily eDiary (UPDD) for the duration of the study

Exclusion Criteria:

* Hypersensitivity to any of the study treatments
* Clearly defined predominant or sole trigger of their chronic urticaria (chronic inducible urticaria)
* Other diseases with symptoms of urticaria or angioedema
* Other skin disease associated with chronic itching that might influence in the investigators opinion the study evaluations and results,
* Known or suspected history of an ongoing, chronic or recurrent infectious disease including but not limited to opportunistic infections (eg tuberculosis, atypical mycobacterioses, listeriosis or aspergillosis), HIV, Hepatitis B/C.
* Pregnant or nursing (lactating) women
* Women of child-bearing potential not using highly effective methods of contraception

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (75):
- United States (11):
  - Novartis Investigative Site, Litchfield Park, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Mission Viejo, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Westminster, California
  - Novartis Investigative Site, Pembroke Pines, Florida
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Ypsilanti, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Grove City, Ohio
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Mendoza, Mendoza Province
  - Novartis Investigative Site, CABA
- Belgium (2):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Liège
- Canada (6):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Niagara Falls, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Verdun, Quebec
  - Novartis Investigative Site, Québec
- Czechia (3):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Prague, Prague 1
  - Novartis Investigative Site, Tábor
- Denmark (2):
  - Novartis Investigative Site, Arhus C
  - Novartis Investigative Site, Copenhagen NV
- France (5):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Rouen
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, München
- Hungary (6):
  - Novartis Investigative Site, Debrecen, Hajdú-Bihar
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Orosháza
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szolnok
- Japan (8):
  - Novartis Investigative Site, Ichinomiya, Aichi-ken
  - Novartis Investigative Site, Funabashi, Chiba
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Koto, Tokyo
  - Novartis Investigative Site, Takaoka, Toyama
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Utrecht
- Poland (5):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Stavropol
- Slovakia (3):
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Svidník
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Madrid
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Denizli
  - Novartis Investigative Site, Talas / Kayseri
- United Kingdom (4):
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Plymouth

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1033

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 311 participants enrolled at 82 investigative sites in 17 countries. This Randomized Set included all randomized subjects, regardless of whether or not they actually received study medication. Subjects were analyzed according to the treatment assigned at randomization.
Pre-assignment Details: Informed consent was obtained from each subject in writing at screening before any study specific procedure was performed. The study was explained to the subject by the investigator or designee, who answered any questions, and written information was also provided.
  Re-screening was allowed once and if a subject was re-screened, then the subject had to sign a new informed consent form.
  .
Groups:
- Placebo Arm: Took matching placebo twice daily
Period: Overall Study
Arm/Group | LOU064 Arm 1 | LOU064 Arm 2 | LOU064 Arm 3 | LOU064 Arm 4 | LOU064 Arm 5 | LOU064 Arm 6 | Placebo Arm
Started | 44 | 44 | 47 | 44 | 44 | 45 | 43
Randomized Set (RAN) | 44 | 44 | 47 | 44 | 44 | 45 | 43
Full Analysis Set (FAS) | 44 | 44 | 47 | 44 | 43 | 45 | 42
Safety Set (SAF) | 44 | 44 | 47 | 44 | 43 | 45 | 42
Completed | 41 | 41 | 45 | 40 | 40 | 36 | 38
Not Completed | 3 | 3 | 2 | 4 | 4 | 9 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 1 | 3 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Technical problems | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0 | 1 | 3
Not completed — Covid-19 pandemic | 0 | 0 | 1 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set included all randomized subjects, regardless of whether or not they actually received study medication. Subjects were analyzed according to the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | LOU064 Arm 1 | LOU064 Arm 2 | LOU064 Arm 3 | LOU064 Arm 4 | LOU064 Arm 5 | LOU064 Arm 6 | Placebo Arm | Total
Number analyzed (Participants) | 44 | 44 | 47 | 44 | 44 | 45 | 43 | 311
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 39 | 44 | 39 | 39 | 41 | 36 | 279
  >=65 years | 3 | 5 | 3 | 5 | 5 | 4 | 7 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (16.04) | 44.0 (16.47) | 45.2 (13.40) | 46.1 (15.21) | 47.4 (14.62) | 44.9 (13.76) | 45.1 (15.24) | 45.0 (14.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 30 | 39 | 32 | 32 | 29 | 25 | 222
  Male | 9 | 14 | 8 | 12 | 12 | 16 | 18 | 89
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 36 | 37 | 40 | 36 | 36 | 36 | 35 | 256
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Asian | 7 | 6 | 7 | 7 | 7 | 9 | 7 | 50
  Native Hawaiian or Other Pacific | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Multiple | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Urticaria Activity Score (UAS7) at Week 4
Description: UAS7 score change (LS mean Change) from baseline at Week 4 estimated with a mixed-effect repeated measurement analysis of UAS7 score change from baseline (FAS)
  The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. The maximum UAS7 value is 42. A higher score indicates worse disease. A negative change score (week 4 score minus Baseline score) indicates improvement.
Time Frame: Baseline, Week 4
Population: Full Analysis Set (FAS) included all randomized subjects. Following intent-to-treat principle, subjects were analyzed according to the treatment and strata assigned to at randomization.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- LOU064 Arm 1: 10 mg LOU064 q.d. capsule once daily
- LOU064 Arm 2: 35 mg capsule q.d. LOU064 once daily
- LOU064 Arm 3: 100 mg capsule q.d. LOU064 once daily
Arm/Group | LOU064 Arm 1 | LOU064 Arm 2 | LOU064 Arm 3 | LOU064 Arm 4 | LOU064 Arm 5 | LOU064 Arm 6 | Placebo Arm
Number analyzed (Participants) | 44 | 44 | 47 | 44 | 43 | 45 | 42
Scores on a scale | -19.10 (1.686) | -19.08 (1.690) | -14.65 (1.624) | -15.99 (1.686) | -20.02 (1.708) | -18.06 (1.691) | -5.44 (1.739)
Statistical Analysis 1: Comparison: LOU064 Arm 1 vs Placebo Arm; Test type: Superiority — LOU064 10 mg q.d; p < 0.0001, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -13.66, 90% CI 2-sided [-17.51 to -9.81], Standard Error of Mean 2.334
Statistical Analysis 2: Comparison: LOU064 Arm 2 vs Placebo Arm; Test type: Superiority — LOU064 35 mg q.d; p < 0.0001, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -13.64, 90% CI 2-sided [-17.49 to -9.78], Standard Error of Mean 2.336
Statistical Analysis 3: Comparison: LOU064 Arm 3 vs Placebo Arm; Test type: Superiority — LOU064 100 mg q.d; p < 0.0001, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -9.21, 90% CI 2-sided [-12.97 to -5.45], Standard Error of Mean 2.277
Statistical Analysis 4: Comparison: LOU064 Arm 4 vs Placebo Arm; Test type: Superiority — LOU064 10 mg b.i.d; p < 0.0001, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -10.55, 90% CI 2-sided [-14.38 to -6.72], Standard Error of Mean 2.319
Statistical Analysis 5: Comparison: LOU064 Arm 5 vs Placebo Arm; Test type: Superiority — LOU064 25 mg b.i.d; p < 0.0001, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -14.58, 90% CI 2-sided [-18.43 to -10.73], Standard Error of Mean 2.334
Statistical Analysis 6: Comparison: LOU064 Arm 6 vs Placebo Arm; Test type: Superiority — LOU064 100 mg b.i.d; p < 0.0001, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -12.62, 90% CI 2-sided [-16.45 to -8.78], Standard Error of Mean 2.327

2. Secondary Outcome: Change From Baseline in Weekly Urticaria Activity Score (UAS7) at Week 12
Description: UAS7 score change (LS mean Change) from baseline at Week 12 estimated with a mixed-effect repeated measurement analysis of UAS7 score change from baseline (FAS)
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | LOU064 Arm 1 | LOU064 Arm 2 | LOU064 Arm 3 | LOU064 Arm 4 | LOU064 Arm 5 | LOU064 Arm 6 | Placebo Arm
Number analyzed (Participants) | 41 | 41 | 45 | 40 | 39 | 35 | 39
Score | -18.11 (1.934) | -17.97 (1.934) | -15.27 (1.850) | -17.67 (1.939) | -20.21 (1.964) | -17.38 (1.985) | -7.87 (2.001)
Statistical Analysis 1: Comparison: LOU064 Arm 1 vs Placebo Arm; Test type: Superiority — LOU064 10 mg q.d; p < 0.0001, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -10.24, 90% CI 2-sided [-14.72 to -5.77], Standard Error of Mean 2.710
Statistical Analysis 2: Comparison: LOU064 Arm 2 vs Placebo Arm; Test type: Superiority — LOU064 35 mg q.d; p = 0.0001, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -10.11, 90% CI 2-sided [-14.58 to -5.63], Standard Error of Mean 2.711
Statistical Analysis 3: Comparison: LOU064 Arm 3 vs Placebo Arm; Test type: Superiority — LOU064 100 mg q.d; p = 0.0027, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -7.40, 90% CI 2-sided [-11.75 to -3.05], Standard Error of Mean 2.635
Statistical Analysis 4: Comparison: LOU064 Arm 4 vs Placebo Arm; Test type: Superiority — LOU064 10 mg b.i.d; p = 0.0002, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -9.80, 90% CI 2-sided [-14.25 to -5.35], Standard Error of Mean 2.696
Statistical Analysis 5: Comparison: LOU064 Arm 5 vs Placebo Arm; Test type: Superiority — LOU064 25 mg b.i.d; p < 0.0001, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -12.35, 90% CI 2-sided [-16.82 to -7.87], Standard Error of Mean 2.714
Statistical Analysis 6: Comparison: LOU064 Arm 6 vs Placebo Arm; Test type: Superiority — LOU064 100 mg b.i.d; p = 0.0003, Mixed Models Analysis; Treatment contrast in LS mean (Change); LS Mean = -9.52, 90% CI 2-sided [-14.03 to -5.01], Standard Error of Mean 2.733

3. Secondary Outcome: Percentage of Participants With Either Complete Absence of Hives and Itch (UAS7=0) or Well-controlled Disease (UAS7<=6)
Description: UAS7=0 and UAS7<=6 response rate over time by treatment group (non-responder imputation) The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. The maximum UAS7 value is 42. A higher score indicates more severe disease. A negative change score (week 4 score minus Baseline score) indicates improvement.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percent of participants
Arm/Group | LOU064 Arm 1 | LOU064 Arm 2 | LOU064 Arm 3 | LOU064 Arm 4 | LOU064 Arm 5 | LOU064 Arm 6 | Placebo Arm
Number analyzed (Participants) | 44 | 44 | 47 | 44 | 43 | 45 | 42
Percent of participants
  UAS7=0 | 29.5 [18.7 to 43.0] | 29.5 [18.7 to 43.0] | 29.8 [19.3 to 42.7] | 31.8 [20.6 to 45.3] | 41.9 [29.3 to 55.5] | 26.7 [16.5 to 39.8] | 14.3 [6.7 to 26.7]
  UAS<=6 | 47.7 [34.8 to 61.0] | 52.3 [39.0 to 65.2] | 38.3 [34.8 to 61.0] | 47.7 [26.6 to 61.0] | 55.8 [42.3 to 68.6] | 42.2 [29.9 to 55.5] | 28.6 [17.7 to 42.3]

4. Secondary Outcome: Cumulative Number of Weeks With an AAS7=0 Response
Description: The Weekly angioedema activity score (AAS) is a validated tool to assess occurrence of episodes of angioedema. If the subject reports the occurrence of angioedema ("opening question") with "no", AAS score for this day is 0. If "yes" is the answer to the opening question, the subject will continue to answer questions about the duration, severity and impact on daily functioning and appearance of the angioedema. The AAS7 is a weekly AAS score (AAS7). Minimum and maximum possible AAS7 scores are 0-105. Higher score means more severe disease.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | LOU064 Arm 1 | LOU064 Arm 2 | LOU064 Arm 3 | LOU064 Arm 4 | LOU064 Arm 5 | LOU064 Arm 6 | Placebo Arm
Number analyzed (Participants) | 44 | 44 | 47 | 44 | 43 | 45 | 42
Weeks | 10.2 (2.33) | 10.5 (2.59) | 10.0 (3.06) | 9.8 (3.05) | 10.3 (2.45) | 9.2 (3.38) | 8.2 (3.50)

5. Secondary Outcome: Percentage of Participants With DLQI Score of 0 or 1
Description: Percentage of subjects with DLQI 0/1 response by treatment group and visit (non-responder imputation)
  The Dermatology Life Quality Index (DLQI) is a 10-item dermatology-specific quality of life (QoL) measure. Subjects rate their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives thinking about the previous 7 days. An overall score is calculated and ranges from 0 to 30 (higher score meaning worse disease-related QoL). A DLQI score of 0 or 1 means that there is no impact of a skin disease on the patient's life.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | LOU064 Arm 1 | LOU064 Arm 2 | LOU064 Arm 3 | LOU064 Arm 4 | LOU064 Arm 5 | LOU064 Arm 6 | Placebo Arm
Number analyzed (Participants) | 44 | 44 | 47 | 44 | 43 | 45 | 42
Percentage of participants
  Week 4 | 38.6 [26.5 to 52.2] | 29.5 [18.7 to 43.0] | 29.8 [19.3 to 42.7] | 29.5 [18.7 to 43.0] | 51.2 [37.8 to 64.3] | 33.3 [22.1 to 46.7] | 16.7 [8.4 to 29.4]
  Week 12 | 34.1 [22.6 to 47.6] | 40.9 [28.6 to 54.4] | 38.3 [26.6 to 51.4] | 40.9 [28.6 to 54.4] | 53.5 [40.0 to 66.5] | 35.6 [24.0 to 48.9] | 28.6 [17.7 to 42.3]

6. Secondary Outcome: Mean Change From Baseline in DLQI Score
Description: Summary of DLQI score and change from baseline
  The Dermatology Life Quality Index (DLQI) is a 10-item dermatology-specific quality of life (QoL) measure. Subjects rate their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives thinking about the previous 7 days. An overall score is calculated and ranges from 0 to 30 (higher score meaning worse disease-related QoL).
Time Frame: Baseline, Week 4 and Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LOU064 Arm 1 | LOU064 Arm 2 | LOU064 Arm 3 | LOU064 Arm 4 | LOU064 Arm 5 | LOU064 Arm 6 | Placebo Arm
Number analyzed (Participants) | 44 | 44 | 47 | 44 | 43 | 45 | 42
Scores on a scale
  Week 4: number analyzed (Participants) | 40 | 42 | 44 | 41 | 39 | 33 | 40
  Week 4 | -9.60 (7.214) | -8.38 (7.241) | -7.18 (7.534) | -6.20 (6.416) | -9.21 (7.994) | -6.15 (5.149) | -3.33 (8.090)
  Week 12: number analyzed (Participants) | 37 | 36 | 40 | 40 | 36 | 33 | 37
  Week 12 | -9.03 (6.216) | -7.31 (9.392) | -6.60 (7.798) | -8.25 (6.551) | -8.97 (8.891) | -6.27 (5.513) | -4.38 (6.780)

7. Secondary Outcome: Area Under the Blood Concentration-time Curve (AUC) of LOU064
Description: Assessment of the area under the blood concentration-time curve (AUC) up to four hours following oral administration at Week 4 and Week 12 .
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | LOU064 Arm 1 | LOU064 Arm 2 | LOU064 Arm 3 | LOU064 Arm 4 | LOU064 Arm 5 | LOU064 Arm 6
Number analyzed (Participants) | 44 | 44 | 47 | 44 | 43 | 45
hr*ng/mL
  Week 4: number analyzed (Participants) | 32 | 30 | 30 | 35 | 32 | 28
  Week 4 | 45.2 (18.4) | 131 (65.4) | 427 (314) | 55.9 (32.3) | 107 (56.8) | 418 (246)
  Week 12: number analyzed (Participants) | 33 | 28 | 29 | 34 | 29 | 24
  Week 12 | 41.8 (19.5) | 159 (151) | 441 (313) | 54.4 (29.4) | 118 (66.6) | 469 (240)

8. Secondary Outcome: Observed Maximum Blood Concentration (Cmax) of LOU064
Description: Assessment of the observed maximum blood concentration (Cmax) of LOU064 following drug administration at Week 4 and Week 12 .
Time Frame: Week 4 and Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LOU064 Arm 1 | LOU064 Arm 2 | LOU064 Arm 3 | LOU064 Arm 4 | LOU064 Arm 5 | LOU064 Arm 6
Number analyzed (Participants) | 44 | 44 | 47 | 44 | 43 | 45
ng/mL
  Week 4: number analyzed (Participants) | 32 | 30 | 30 | 35 | 32 | 28
  Week 4 | 27.6 (13.7) | 67.2 (32.7) | 194 (142) | 32.2 (18.7) | 55.5 (34.7) | 196 (144)
  Week 12: number analyzed (Participants) | 33 | 28 | 29 | 35 | 29 | 25
  Week 12 | 26.1 (14.5) | 80.3 (53.9) | 199 (137) | 31.2 (16.0) | 64.9 (42.3) | 219 (125)

9. Secondary Outcome: Time to Reach the Maximum Concentration (Tmax) of LOU064
Description: Assessment of the time to reach the maximum concentration (Tmax) of LOU064 following drug administration at Weeks 4 and 12
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | LOU064 Arm 1 | LOU064 Arm 2 | LOU064 Arm 3 | LOU064 Arm 4 | LOU064 Arm 5 | LOU064 Arm 6
Number analyzed (Participants) | 44 | 44 | 47 | 44 | 43 | 45
hours
  Week 4: number analyzed (Participants) | 32 | 30 | 30 | 35 | 32 | 28
  Week 4 | 1.33 [0.00 to 4.00] | 1.54 [0.00 to 4.00] | 1.52 [0.500 to 3.00] | 0.900 [0.00 to 2.00] | 1.15 [0.00 to 3.02] | 1.52 [0.00 to 3.08]
  Week 12: number analyzed (Participants) | 33 | 28 | 29 | 35 | 29 | 25
  Week 12 | 1.17 [0.00 to 4.08] | 1.48 [0.500 to 4.00] | 1.61 [0.00 to 4.00] | 1.17 [0.500 to 4.00] | 1.32 [0.00 to 4.00] | 1.39 [0.5000 to 4.00]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events were collected after signature of the informed consent form until 30 days after last dose of study treatment, and up to 16 weeks
Description: AEs and SAEs are any untoward sign or symptom that occurs during the study treatment and up to 16 weeks
Groups:
- LOU064 10mg q.d.: 10 mg LOU064 qd capsule once daily
- LOU064 35mg q.d.: 35 mg capsule qd LOU064 once daily
- LOU064 100mg q.d.: 100 mg capsule qd LOU064 once daily
- LOU064 10mg b.i.d.: 10 mg capsule LOU064 bid
- LOU064 25mg b.i.d.: 25 mg capsule LOU064 bid
- LOU064 100mg b.i.d.: 100 mg capsule LOU064 bid
- Any LOU064: Any LOU064
- Placebo: Participants took matching placebo twice daily
Arm/Group | LOU064 10mg q.d. | LOU064 35mg q.d. | LOU064 100mg q.d. | LOU064 10mg b.i.d. | LOU064 25mg b.i.d. | LOU064 100mg b.i.d. | Any LOU064 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44 | 0/47 | 0/44 | 0/43 | 0/45 | 0/267 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/44 | 0/47 | 2/44 | 2/43 | 0/45 | 5/267 | 0/42
Other Adverse Events (participants affected / at risk) | 15/44 | 13/44 | 10/47 | 12/44 | 11/43 | 13/45 | 74/267 | 11/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LOU064 10mg q.d. (N=44) | LOU064 35mg q.d. (N=44) | LOU064 100mg q.d. (N=47) | LOU064 10mg b.i.d. (N=44) | LOU064 25mg b.i.d. (N=43) | LOU064 100mg b.i.d. (N=45) | Any LOU064 (N=267) | Placebo (N=42)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LOU064 10mg q.d. (N=44) | LOU064 35mg q.d. (N=44) | LOU064 100mg q.d. (N=47) | LOU064 10mg b.i.d. (N=44) | LOU064 25mg b.i.d. (N=43) | LOU064 100mg b.i.d. (N=45) | Any LOU064 (N=267) | Placebo (N=42)
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 4 | 0 | 1 | 7 | 2
Nausea (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 1 | 2 | 10 | 0
Pyrexia (General disorders) | 3 | 0 | 0 | 2 | 1 | 0 | 6 | 0
Nasopharyngitis (Infections and infestations) | 7 | 2 | 2 | 4 | 4 | 4 | 23 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2 | 0 | 3 | 0 | 8 | 1
Headache (Nervous system disorders) | 1 | 7 | 4 | 3 | 6 | 5 | 26 | 6
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 4 | 2 | 2 | 16 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT03926611/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT03926611/SAP_001.pdf